CLINICAL TRIAL: NCT01139255
Title: The Use of Podcasting and Mobile Media to Promote Weight Loss and Increase Fruit and Vegetable Intake Among Overweight Adults
Brief Title: Pounds Off Digitally (POD): The Use of Podcasting and Mobile Media to Promote Weight Loss
Acronym: POD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Brie Turner-McGrievy, UNC Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0930
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-06

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Podcasting + mobile media (Experimental)
  Interventions: Behavioral: Podcasting + mobile media
- Podcasting (Active Comparator)
  Interventions: Behavioral: Podcasting + mobile media

INTERVENTIONS:
Behavioral: Podcasting + mobile media — Use of a weight loss podcast designed with health behavior theory

SUMMARY:
Overweight and obesity play a role in both cancer incidence and survival rates. Many people have found attending weight loss support groups to be time-intensive. Past research has shown electronic media, particularly the Web, to be effective in producing weight loss. The Web, however, lacks portability, which prevents people from accessing the information when it is convenient for them. Providing weight loss information via podcasting (audio files that may be listened to on portable audio players) may allow people to receive weight loss tips anywhere. A previous research study showed that podcasts emphasizing healthy eating and exercise can help people lose weight. This study was short-term and did not include additional social support. The purpose of this research project is to assess the effectiveness of a weight loss intervention delivered through podcasts as compared to the same podcast with added mobile media such as self-monitoring software (such as a pedometer) and support delivered via a social networking site. For this research study, the investigators will conduct a 6-month study in 104 overweight adults to determine if a podcast plus mobile media support leads to greater weight loss than a podcast alone.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18-60 years old
* be a non-smoker
* live in the Chapel Hill, NC area
* be able to attend monitoring visits at baseline, 3-months, and 6-months
* have access to the Internet and a computer
* have access to an Internet-capable mobile device (such as an iPhone, iPod Touch, or Blackberry) and an MP3 player (this may be the same device)
* have access to a scale for self-monitoring weight
* be willing to be randomized to either group
* be free of psychiatric diseases, drug or alcohol dependency, or uncontrolled thyroid conditions
* be free of major health conditions, such as heart conditions, diabetes, and past incidence of stroke
* have MD consent for participation if currently on blood pressure medications, have issues with dizziness, or have bone or joint issues.
* able to prepare all their own meals (i.e. not living on-campus)

Exclusion Criteria:

* should not be pregnant, anticipating on becoming pregnant in the next 7 months, or currently breastfeeding
* be free of an eating disorder as screened by the Eating disorder Screen for Primary care [ESP].
* no current participation in a weight loss program or taking weight loss medications (although participants may be trying to lose weight on their own)
* have not participated in previous podcasting weight loss research

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2010-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Weight loss | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Brie Turner-McGrievy, PhD, MS, RD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC-Chapel Hill Weight Research Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Turner-McGrievy G, Tate D. Tweets, Apps, and Pods: Results of the 6-month Mobile Pounds Off Digitally (Mobile POD) randomized weight-loss intervention among adults. J Med Internet Res. 2011 Dec 20;13(4):e120. doi: 10.2196/jmir.1841. PMID 22186428
- See also: Related Info — http://www.uncweightresearch.org/